CLINICAL TRIAL: NCT00779311
Title: A Phase I Trial Evaluating mFOLFOX6 and Avastin With Nexavar as First-Line Treatment for Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Dose limiting toxicity at the lowest planned dose level.
Sponsor: Accelerated Community Oncology Research Network (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFMSMCRC0706
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Results first posted 2011-10-26 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Sorafenib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimenal (Experimental): All eligible patients will receive the mFOLFOX6 regimen at full dose followed by IV bevacizumab 5mg/kg on Day 1 of each treatment cycle. Sorafenib will be administered daily throughout treatment beginning on day 1
  Interventions: Drug: sorafenib; Drug: bevacizumab; Drug: mFOLFOX6 regimen

INTERVENTIONS:
Drug: sorafenib — Sorafenib will be administered daily starting day 1 at 200mg QOD at Dose Level 1; 200mg/day at Dose Level 2; 200mg BID (5 days on/ 2 days off) at Dose Level 3; 200mg BID at Dose Level 4; and 400mg BID at Dose Level 5.
  Other Names: Nexavar
Drug: bevacizumab — Bevacizumab will be administered as 5mg/kg IV on Day 1 of each treatment cycle.
  Other Names: Avastin
Drug: mFOLFOX6 regimen — The mFOLFOX6 regimen will be administered on Day 1 of each treatment cycle. This regimen consists of oxaliplatin 85 mg/m2 IV given over 2 hours, leucovorin 400 mg/m2 IV given over 2 hours, and fluorouracil 400 mg/m2 IV bolus, followed by fluorouracil 1200 mg/m2 per day for 2 days continuous infusion.

SUMMARY:
This research study is being performed at approximately 3 sites associated with Accelerated Community Oncology Research Network, Inc. (ACORN). Approximately 45 subjects will take part in this study.

In this study, everyone will receive the same dose of mFOLFOX6 and Avastin. There will be five groups of subjects. Each group of subjects will receive a higher dose of Nexavar than the previous group. This will continue until a subject group has a major side effects from the dose they are given. This is so that the sponsor can determine the highest dose of Nexavar that can be used with mFOLFOX6 and AVastin (this is called the maximum tolerated dose or MTD).

DETAILED DESCRIPTION:
This is an investigator-initiated, multicenter, network, Phase 1, open-label, dose-ranging study. The maximum sample size will be 45 patients (up to 30 patients for determining MTD at Phase I, and an additional 15 patients to provide for estimate of progression free survival). All eligible patients will receive the mFOLFOX6 regimen at full dose followed by IV bevacizumab 5mg/kg on Day 1 of each treatment cycle. Treatment cycle length is 2 weeks (Q2W). Sorafenib will be administered daily throughout treatment beginning on day 1.

Dose limiting toxicity will be defined as any grade 4 hematologic event or any grade 3 or 4 non-hematologic event occurring during cycle 1 or 2 that is attributable to sorafenib or the combination. The following events are excluded from this definition: grade 3 nausea and/or vomiting responsive to antiemetics; grade 3 fever or infection; grade 3 diarrhea responsive to antidiarrheal therapy.

Three patients will be enrolled at a dose level and observed for dose-limiting toxicities (DLTs) for 2 cycles of treatment. Dose escalation for sorafenib will depend on the number of patients experiencing DLT(s) as follows:

* If 0/3 patients experience DLT(s), then 3 more patients are treated at the next higher dose.
* If 1/3 patients experiences DLT(s), then 3 more patients are enrolled at that dose. If 1/6 of the patients treated at that dose experiences DLT(s), then the next cohort is treated at the next higher dose. However, if ≥2/6 patients experience DLT(s) at that dose, then the MTD is considered to have been exceeded. At that point, 3 more patients are treated at the next lower dose, unless 6 have already been treated at that lower dose.
* If ≥2/3 patients experience DLT(s) at a dose, then 3 more patients are enrolled at the next lower dose unless 6 patients have already been treated at that dose.

Dose escalation will continue until the MTD is determined or until all dose levels have been completed. The MTD is defined as the dose at which ≤1 of 6 patients experience DLT(s), and above which ≥2 of 6 patients experience DLT(s). If the MTD is at Dose Level 2 (or lower), then the study will be terminated and no further patients will be enrolled.

Once the MTD for sorafenib combined with mFOLFOX6 and bevacizumab has been determined, an additional 15 patients with mCRC will be enrolled into an extension of the Phase 1 study. These patients will be treated at the MTD for sorafenib with the combination therapy to assess PFS and safety of the regimen as first-line therapy in mCRC. All patients will be eligible for indefinite treatment in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* No prior chemotherapy for metastatic disease.
* Histologically proven colorectal carcinoma.
* Measurable disease by RECIST criteria.
* Age: at least 18 years.
* ECOG performance status of 0 or 1 at study entry.
* Adequate bone marrow, liver and renal function at study entry as assessed by the following:

  * Hemoglobin >9.0 g/dL.
  * ANC ≥1500/mm3.
  * Platelet count ≥100,000/mm3.
  * Total bilirubin ≤1.5 times x ULN.
  * ALT and AST ≤2.5 × ULN (≤5 × ULN for patients with liver involvement).
  * Creatinine ≤1.5 × ULN.
* INR <1.5 or a PT/PTT within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate after discussion with ACORN. For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.
* Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to the start of treatment.
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Patients should use adequate birth control for at least 3 months after the last administration of sorafenib.
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.

Exclusion Criteria:

* Prior use of bevacizumab.
* Neuropathy ≥ Grade 2 per CTCAE v3.0.
* Diarrhea ≥ Grade 2 per CTCAE v3.0 within 4 weeks of study treatment start.
* ECOG performance status ≥ 2.
* Proteinuria at baseline: patients discovered to have > 2+ proteinuria at baseline should undergo a 24 hour urine collection and must demonstrate < 1 gram of protein in 24 hours to be eligible.
* Active malignancy other than mCRC (except non-melanoma skin cancer; in situ carcinoma of the cervix; in situ carcinoma of the breast) within the last 5 years.
* Treatment with radiotherapy within 2 weeks of enrollment.
* Cardiac disease: Congestive heart failure > Class II NYHA. Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Known brain metastasis. Patients with neurological symptoms must undergo a CT scan/ MRI of the brain to exclude brain metastasis.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mm Hg or diastolic pressure > 90 mm Hg, despite optimal medical management.
* Known human immunodeficiency virus infection or chronic Hepatitis B or C.
* Active clinically serious infection > Grade 2 per CTCAE v3.0.
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Pulmonary hemorrhage/bleeding event ≥ Grade 2 per CTCAE v3.0 within 4 weeks of study treatment start.
* Any other hemorrhage/bleeding event ≥ Grade 3 per CTCAE v3.0 within 4 weeks of study treatment start.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of bleeding diathesis or coagulopathy.
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of study treatment start; fine needle aspiration or central venous line placement for chemotherapy administration within 7 days of study treatment start.
* Use of daily corticosteroids, St. John's Wort, rifampin (rifampicin), phenytoin, carbamazepine, phenobarbital, ketoconazole. Dexamethasone may only be used as an antiemetic or as a premedication for a bevacizumab hypersensitivity reaction during participation in this study.
* Known or suspected allergy to sorafenib or any other agent given in the course of this trial.
* Any condition that impairs patient's ability to swallow whole pills.
* Any malabsorption problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Schnell, MD, Principal Investigator — Central Georgia Cancer Care
Locations (3):
- United States (3):
  - Central Georgia Cancer Care, Macon, Georgia
  - Hematology Oncology Centers of the Northern Rockies, Billings, Montana
  - The West Clinic, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three community oncology research sites across the US within the ACORN Network participated in this study. Enrollment started in October 2008 and was closed early in April 2010 due to two subjects experiencing DLT at the lowest dose level.
Pre-assignment Details: Informed consent was obtained from all subjects. All subjects underwent a screening period that could last up to 4 weeks during which pre-study assessments were completed. All subjects received mFOLFOX6, bevacizumab, and sorafenib. Subjects were assigned to a Dosage Level at the time of enrollment.
Groups:
- Dose Level (DL) 1 for MTD Determination: All eligible patients will receive the mFOLFOX6 regimen at full dose followed by IV bevacizumab 5mg/kg on Day 1 of each treatment cycle, and sorafenib 200mg every other day.
- Dose Level (DL) 2 for MTD Determination: All eligible patients will receive the mFOLFOX6 regimen at full dose followed by IV bevacizumab 5mg/kg on Day 1 of each treatment cycle, and sorafenib 200mg every day.
- Dose Level (DL) 3 for MTD Determination: All eligible patients will receive the mFOLFOX6 regimen at full dose followed by IV bevacizumab 5mg/kg on Day 1 of each treatment cycle, and sorafenib 200mg twice a day, 5 days on followed by 2 days off.
- Dose Level (DL) 4 for MTD Determination: All eligible patients will receive the mFOLFOX6 regimen at full dose followed by IV bevacizumab 5mg/kg on Day 1 of each treatment cycle, and sorafenib 200mg twice a day.
- Dose Level (DL) 5 for MTD Determination: All eligible patients will receive the mFOLFOX6 regimen at full dose followed by IV bevacizumab 5mg/kg on Day 1 of each treatment cycle, and sorafenib 400mg twice a day.
Period: Overall Study
Arm/Group | Dose Level (DL) 1 for MTD Determination | Dose Level (DL) 2 for MTD Determination | Dose Level (DL) 3 for MTD Determination | Dose Level (DL) 4 for MTD Determination | Dose Level (DL) 5 for MTD Determination
Started | 8 (2 of 6 patients were not evaluable for DLT assessment and were replaced for a total of 8 enrolled.) | 0 | 0 | 0 | 0
Dose Limiting Toxicity (DLT) Evaluation | 6 | 0 | 0 | 0 | 0
Completed | 8 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level (DL) 1 for MTD Determination | Dose Level (DL) 2 for MTD Determination | Dose Level (DL) 3 for MTD Determination | Dose Level (DL) 4 for MTD Determination | Dose Level (DL) 5 for MTD Determination | Total
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0 | 8
Age Categorical [Number; unit: participants]
  <=18 years | 0 |  |  |  |  | 0
  Between 18 and 65 years | 3 |  |  |  |  | 3
  >=65 years | 5 |  |  |  |  | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 62.0 (11.40) |  |  |  |  | 62.0 (11.40)
Gender [Number; unit: participants]
  Female | 3 |  |  |  |  | 3
  Male | 5 |  |  |  |  | 5
Region of Enrollment [Number; unit: participants]
  United States | 8 |  |  |  |  | 8

OUTCOME MEASURES:

1. Primary Outcome: Determination of the Maximum Tolerated Dose (MTD) of Sorafenib When Given in Combination With mFOLFOX6 and Bevacizumab
Description: The MTD of sorafenib was determined using a standard 3 + 3 dose escalation cohort design. The total sample and the number of patients who receive each dose depends on the frequency of dose limiting toxicities (DLT) at each dosage. If 0 out of 3 patients experience a DLT at a given dosage level, 3 patients will be enrolled at the next dosage level. If greater than or equal to 2 patients experience a DLT at a given dosage level, dosage escalation will be stopped. If 1 out of 3 patients experience a DLT at a given dosage level, 3 patients are enrolled at the same dosage level.
Time Frame: MTD was assessed during the first 2 cycles of treatment (i.e., the first 4 weeks of treatment since cycle length is 2 weeks)
Population: 3 patients (pts) were enrolled at DL 1 with 1/3 experiencing DLT, so 3 additional pts were enrolled at DL 1. 2 of those additional pts were not evaluable for DLT assessment and were replaced. 2 more pts were enrolled for a total of 8 pts, and 1 of these pts experienced a DLT. All of the 8 pts enrolled received sorafenib at DL 1.
Measure: Number; unit: mg every other day
Arm/Group | Dose Level (DL) 1 for MTD Determination | Dose Level (DL) 2 for MTD Determination | Dose Level (DL) 3 for MTD Determination | Dose Level (DL) 4 for MTD Determination | Dose Level (DL) 5 for MTD Determination
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0
mg every other day | 200 |  |  |  |

2. Secondary Outcome: Determination of Progression Free Survival (PFS) Among Patients on This Regimen
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever comes first.
Time Frame: PFS was measured from day 1 of treatment until time of progression (assessed every 8 weeks) or death, whichever came first.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Level (DL) 1 for MTD Determination | Dose Level (DL) 2 for MTD Determination | Dose Level (DL) 3 for MTD Determination | Dose Level (DL) 4 for MTD Determination | Dose Level (DL) 5 for MTD Determination
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0
Months | 10.61 [3.61 to 13.40] |  |  |  |

3. Secondary Outcome: Determination of Quality of Life (QoL) as Indicated by Patient Care Monitor (PCM) Data Among Patients on This Regimen
Description: The subject answers questions from the following 6 categories: general physical symptoms, treatment side effects, distress, despair, impaired performance, and impaired ambulation. Each question has a scale from 0 through 10, where 0 is not a problem and 10 is as bad as possible. The frequency of patient reported severe (rated as >=7) symptoms reported from the set of symptoms assessed by the PCM.
Time Frame: The PCM questionnaire was administered on day 1 of each cycle (approximately every 2 weeks) during study treatment.
Population: The number of patients out of the total sample of 8 patients who reported severe (rated as >=7) symptoms as assessed by the PCM. Symptoms with 0 patients reporting severe symptoms have been omitted.
Measure: Number; unit: Participants
Arm/Group | Dose Level (DL) 1 for MTD Determination | Dose Level (DL) 2 for MTD Determination | Dose Level (DL) 3 for MTD Determination | Dose Level (DL) 4 for MTD Determination | Dose Level (DL) 5 for MTD Determination
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0
Participants
  Fatigue | 3 |  |  |  |
  Change in taste | 2 |  |  |  |
  Mouth sores/ulcers | 1 |  |  |  |
  Sore throat | 1 |  |  |  |
  Trouble swallowing | 1 |  |  |  |
  Day sweat | 1 |  |  |  |
  Night sweat | 1 |  |  |  |
  Reduced sexual enjoyment, interest, or performance | 2 |  |  |  |
  Heartburn | 1 |  |  |  |
  Nausea | 2 |  |  |  |
  Problem with urination | 1 |  |  |  |
  Bruising | 1 |  |  |  |
  New lump/mass | 1 |  |  |  |
  Hair loss | 1 |  |  |  |
  Nails change | 1 |  |  |  |
  Joint pain | 2 |  |  |  |
  Muscle aches | 2 |  |  |  |
  Weakness of body parts | 2 |  |  |  |
  Burning sensation in hands or feet | 2 |  |  |  |
  Numbness/tingling | 2 |  |  |  |
  Trouble sleeping at night | 2 |  |  |  |
  Pain | 1 |  |  |  |
  Attend paid job | 2 |  |  |  |
  Attend social activity | 1 |  |  |  |
  Hard work or activity | 2 |  |  |  |
  Household work | 1 |  |  |  |
  Light work or activity | 1 |  |  |  |
  Run | 2 |  |  |  |
  Walk | 1 |  |  |  |
  Crying/feeling like crying | 1 |  |  |  |
  Feeling helpless | 1 |  |  |  |
  Feeling hopeless | 1 |  |  |  |
  Lost interest in people | 1 |  |  |  |
  Nervous, tense, anxious | 2 |  |  |  |
  Worry | 2 |  |  |  |

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning on day 1 of study treatment until one month after the end of study treatment.
Description: Systematic Assessment - subjects were assessed for adverse events on day 1 of each cycle (every other week) by either the research coordinator, treating physician, or other appropriate sub-investigator.
Arm/Group | Dose Level (DL) 1 for MTD Determination | Dose Level (DL) 2 for MTD Determination | Dose Level (DL) 3 for MTD Determination | Dose Level (DL) 4 for MTD Determination | Dose Level (DL) 5 for MTD Determination
Serious Adverse Events (participants affected / at risk) | 5/8 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 8/8 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level (DL) 1 for MTD Determination (N=8) | Dose Level (DL) 2 for MTD Determination (N=0) | Dose Level (DL) 3 for MTD Determination (N=0) | Dose Level (DL) 4 for MTD Determination (N=0) | Dose Level (DL) 5 for MTD Determination (N=0)
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level (DL) 1 for MTD Determination (N=8) | Dose Level (DL) 2 for MTD Determination (N=0) | Dose Level (DL) 3 for MTD Determination (N=0) | Dose Level (DL) 4 for MTD Determination (N=0) | Dose Level (DL) 5 for MTD Determination (N=0)
Anemia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 2 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 5 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 2 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0 | 0
Temperature intolerance (General disorders) | 3 | 0 | 0 | 0 | 0
Thrombosis in device (General disorders) | 1 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Laryngitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dysesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 4 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 3 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Peripheral coldness (Vascular disorders) | 4 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Early termination due to the MTD determined to be Dose Level 1, leading to a small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication or presentation of Sponsored Research results, Researcher agrees to provide Bayer with such presentation, abstract, or manuscript at least 30 days prior to its presentation or submission for the sole purpose of allowing Bayer to redact Confidential Information and protect any existing or future patents.